CLINICAL TRIAL: NCT00477906
Title: Comparison of M-Vax Plus Low Dose Interleukin-2 Versus Placebo Vaccine Plus Low Dose Interleukin-2 in Patients With Stage IV Melanoma
Brief Title: M-Vax + Low Dose Interleukin-2 Versus Placebo Vaccine in Metastatic Melanoma in Patients With Stage IV Melanoma
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: AVAX Technologies (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: A/100/0402
Record Dates: First submitted 2007-05-22; First posted 2007-05-24 (Estimated); Last update posted 2015-12-03 (Estimated); Status verified 2015-12

CONDITIONS: Melanoma
Keywords: melanoma; vaccine; metastatic; autologous
MeSH Terms: conditions — Melanoma; Neoplasm Metastasis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): MVax + BCG + cyclophosphamide + IL2
  2:1 randomization - MVax:Control
  Interventions: Biological: M-Vax- autologous, hapten-modified melanoma vaccine
- 2 (Placebo Comparator): Placebo Vaccine + BCG + cyclophosphamide + IL2
  Interventions: Biological: M-Vax- autologous, hapten-modified melanoma vaccine

INTERVENTIONS:
Biological: M-Vax- autologous, hapten-modified melanoma vaccine — Autologous, DNP-modified melanoma cells in suspension Dose: 12+-8 million cells Route: intradermal Frequency: weekly X7 + 6 month booster

SUMMARY:
Previous studies suggests that M-Vax, a melanoma vaccine prepared from patients own cancer cells, can stimulated patients' immune system to react against their cancer. AVAX has identified a dose and schedule of administration of M-Vax that work optimally. In this study, AVAX will determine whether M-Vax is effective in shrinkage of melanomas that have spread (stage IV). To increase it effectiveness, M-Vax administration will be followed by administration of low doses of interleukin-2 (IL2), a marketed drug that is known to stimulate immunity and cause some shrinkage of melanomas. Two-thirds of patients will receive M-Vax + IL2, and one-third will receive a placebo vaccine + IL2. The study is blinded so that neither the patients nor their physicians know which material they are receiving.

To be eligible for this study, patients must have at least one melanoma tumor that can be surgically removed and made into a vaccine. In addition, they must have melanoma that has spread to to the lungs or to soft tissue sites (under the skin, on the surface of the skin, lymph nodes). Eligible patients may have previously received one treatment (for example, chemotherapy) for their melanoma.

Side effects of M-Vax are expected to be mild; the most common is the development of sore pimples at the site of vaccine injections. The low dose IL2 may cause some fatigue and other mild symptoms.

It is expected that 387 patients will be treated in this study.

DETAILED DESCRIPTION:
M-Vax is a therapeutic melanoma vaccine consisting of autologous melanoma cells that have been irradiated and then modified with the hapten, dinitrophenyl (DNP). There is a large amount of published evidence that hapten modification makes visible to the immune system antigens, including tumor antigens, that otherwise do not elicit an immune response.

This is a Phase III, randomized, placebo-controlled, double-blind, multi-centered trial of M-Vax in patients with stage IV melanoma with measurable metastases in lung and/or soft tissues. To be eligible for screening, patients will have undergone surgery for therapeutic intervention, which yields an adequate amount of melanoma tumor cells for preparation of vaccines, which pass vaccine release testing. Eligible patients who meet all inclusion/exclusion criteria will be enrolled in the study.

Patients will be assigned in a double-blind fashion to M-Vax or Placebo Vaccine at a 2:1 ratio (M-Vax:Placebo Vaccine). The dose of M-Vax will be 4.0-20.0x10(6) DNP-modified autologous melanoma tumor cells. The Placebo Vaccine will consist of diluent only. An initial dose of M Vax or Placebo Vaccine will be administered without BCG followed by low dose cyclophosphamide (300 mg/m2 iv). Then M Vax or Placebo Vaccine mixed with Bacillus of Calmette and Guérin (BCG) will be administered weekly for 6 weeks. Four courses of interleukin-2 (IL2) will be administered to all patients starting about 2 weeks after the last vaccine; each course will consist of 3 million units/m2 subcutaneously daily for 5 days followed by a 16-day rest period.

The primary endpoints of the study are: 1)Best overall anti-tumor response, and 2)Survival, measured by % surviving at two years. Patients will be evaluated for anti-tumor response by modified RECIST criteria between weeks 24 and 25 (i.e., 5-6 weeks after completion of IL2). At the 6-month point patients who remain on study will receive an additional single booster dose of M-Vax or Placebo Vaccine mixed with BCG. This will be followed by four more courses of IL2. Two additional evaluations for anti-tumor response will take place at the 38-39 week (month 9) and one-year points. Then patients will be regularly evaluated for tumor status and adverse events until evidence of tumor progression that requires new therapy. Patients who remain on-study will be followed until death but for a maximum of 5 years.

The intended sample size is 387, and there will be about 25 sites participating in the United States, Europe, and Israel. An interim analysis will be performed after half the patients have been accrued.

ELIGIBILITY:
Inclusion Criteria:

* Stage IV metastatic melanoma of cutaneous or mucosal origin or without known primary site

  * At least one metastatic mass that is surgically resectable, excluding metastases in brain, bowel, or bone
  * Successful preparation of a vaccine that meets quality control release criteria
  * Following surgery for vaccine preparation, subjects must have at least one measurable metastasis defined by modified RECIST criteria. Non-measurable metastases may also be present. Residual metastases (measurable or non-measurable) must be limited to skin (dermal or subcutaneous), lymph node, or lung, or a combination of these.
  * No prior systemic treatment or one prior systemic treatment for metastatic melanoma, not counting post-surgical adjuvant treatment with alpha interferon
  * Minimum of one month and maximum of 4 months since the surgery
  * Expected survival of at least 6 months
  * Karnofsky performance status at least 80
  * Signed informed consent

Exclusion Criteria:

* Failure to prepare a vaccine that meets all quality control release criteria

  * Uveal melanoma
  * Post-surgical residual metastases in sites other than specified in 6.1
  * Brain metastases, current or past (unless successfully treated at least one year prior to enrollment)
  * Hepatic transaminase > 2.5 x ULN
  * Total bilirubin > 2.0 mg/Dl
  * Creatinine > 2.0 mg/Dl
  * Hemoglobin < 10.0 g/Dl
  * WBC < 3,000 /mm3
  * Platelet count < 100,000/mm3
  * Limited field radiotherapy, i.e., limited to recent surgical site, less than 4 weeks prior to first dose of vaccine
  * Major field radiotherapy less than 6 months prior to first dose of vaccine
  * Any systemic treatment for metastatic melanoma, including chemotherapy, cytokines, or investigational drugs less than 2 months prior to first dose of vaccine
  * Previous administration of M-Vax
  * Prior splenectomy
  * Administration of systemic steroids less than 4 weeks prior to first dose of vaccine. Topical steroids are allowed during the study, provided these are not applied to vaccine injection sites. Inhaled aerosol steroids also are allowed during the study.
  * Administration of immunosuppressive drugs less than 4 weeks prior to first dose of vaccine
  * Administration of antitubercular drugs (e.g., isoniazid, rifampin, streptomycin) less than 4 weeks prior to first dose of vaccine
  * HIV 1/2 positive by ELISA, confirmed by Western blot
  * Hepatitis B surface antigen or hepatitis C antibody positive
  * Other malignancy within 5 years except: curatively treated non-invasive melanoma, non-melanomatous skin cancer, carcinoma in situ of the uterine cervix, or early stage (stage A or B1) prostate cancer
  * Autoimmune diseases that would interfere with an immunologic response (e.g., systemic lupus erythematosus, multiple sclerosis or ankylosing spondylitis)
  * Concurrent medical condition that would preclude compliance or immunologic response to study treatment
  * Concurrent serious infection, including active tuberculosis, or other serious medical condition
  * Pregnancy or lactation (serum human chorionic gonadotropin [HCG] test must be negative in fertile women at screening visit)
  * Known gentamicin allergy
  * Anergic, defined by the inability to make a DTH to at least one of the following: candida, mumps, tetanus or trichophyton (based upon availability)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 387 (Estimated)
Dates: Start 2016-07; Primary Completion 2019-01 (Estimated); Study Completion 2021-01 (Estimated)

PRIMARY OUTCOMES:
Best overall anti-tumor response. | 1 year
Survival - % patients surviving at two years | 2 years

SECONDARY OUTCOMES:
Safety | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Henry E Schea, Study Director — AVAX Technologies

REFERENCES:
- [Background] Berd D, Sato T, Maguire HC Jr, Kairys J, Mastrangelo MJ. Immunopharmacologic analysis of an autologous, hapten-modified human melanoma vaccine. J Clin Oncol. 2004 Feb 1;22(3):403-15. doi: 10.1200/JCO.2004.06.043. Epub 2003 Dec 22. PMID 14691123
- [Result] Berd D, Sato T, Cohn H, Maguire HC Jr, Mastrangelo MJ. Treatment of metastatic melanoma with autologous, hapten-modified melanoma vaccine: regression of pulmonary metastases. Int J Cancer. 2001 Nov;94(4):531-9. doi: 10.1002/ijc.1506.abs. PMID 11745440